

Impact of Maxillomandibular Advancement Upon the Pharyngeal Airway Volume and the Apnea-hypopnea Index in the Treatment of Obstructive Sleep Apnea.

## INFORM CONSENT VERSION 1.0 OCTOBER 30, 2017

**RUNNING TITLE:** OSAS-OS - Maxillomandibular Advancement in the Treatment of Obstructive Sleep Apnea

NCT No: NCT03796078



## Anexo 4

| Main Researcher: Hernández-Alfaro F. | |
|---|---|
| secondary researchers: Giralt-Hernando M, Valls-Ontañón A. Title: Impact of Maxillomandibular Advancement Upon the Pharyngeal Airway Volume and the Apnea-hypopnea Index in the Treatment of Obstructive Sleep Apnea. NCT: NCT03796078 | |
| this consent form, which complies with the pro<br>December 13, on Personal Data Protection (L | me. questions to the responsible professional. d understand that my participation is entirely vithout affecting my future medical care. By to my personal data being used as described in |
| Patient's signature | Date |
| D number | |
| STATEMENT OF THE INVESTIGATOR | |
| The patient who signs this consent form has received detailed oral and written information from the professional about the process and nature of this research study and has had the opportunity to ask any questions regarding the nature, risks and benefits of their participation in this study. | |
| nvestigator's signature | Date |

## **INFORMED CONSENT**



Dr Hernández-Alfaro